CLINICAL TRIAL: NCT05694104
Title: China Nutrition Fundamental Data 2020
Acronym: CNFD 2020
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: National Institute of Hospital Administration, National Health Commission (Unknown)
Responsible Party: Principal Investigator, Wei Chen, Professor, Peking Union Medical College Hospital
Other Study IDs: ZS-2614
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Nutritional Status of Chinese Inpatients；Nutritional Service Capacity of Medical Institutions in China

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Malnutrition — For the diagnosis of malnutrition, we adopted the Global Leadership Initiative on Malnutrition (GLIM) scheme based on three phenotypic criteria (non-volitional weight loss, low body mass index, and reduced muscle mass) and two etiologic criteria (reduced food intake or assimilation, and inflammation or disease burden). To diagnose malnutrition at least one phenotypic criterion and one etiologic criterion should be present in patients with nutritional risk.

SUMMARY:
Malnutrition caused by reduced food intake or assimilation and varying degrees of acute or chronic inflammation is a serious and underappreciated risk factor for adverse clinical outcomes. Despite the substantial health and economic burden, malnutrition remains to affect a considerable proportion of hospitalized patients worldwide. Nationally representative studies from the USA, Australia, and European countries have reported prevalence figures in the range of 8.9% to 80.4%. However, national data in some resource-poor countries, such as China, the largest developing country in the world, are scarce.

We did the China Nutrition Fundamental Data 2020 in a large, nationally representative sample of Chinese adult inpatients to 1) Explore the relationship between nutrition and health; 2) Understand the capacity of nutrition services in Chinese medical institutions.

This project adopted a multistage, stratified, cluster-sampling procedure based on administrative divisions in China. For each participant, a structured interview was done by trained nutritionists or clinicians. The following data were acquired: weight change within and beyond six months, food intake change within two weeks, nutrition therapy during this hospitalization, and laboratory tests. We also collected information on participants' sociodemographic characteristics and medical history. We took physical measurements, including height, weight, waist circumference, hip circumference, mid-arm circumference, calf circumference, handgrip strength, and blood pressure following standard protocols. Body composition was measured using bioimpedance analysis (BIA). In total, 54677 inpatients from 291 project hospitals completed information collection.

In addition, we collected information on the number of beds, the nutrition support team, the nutrition treatment plan and the construction of a full-time nutrition physician or nutrition nurse, the routine monitoring methods, interventions, and distribution of brochures for patients with malnutrition or nutritional risk in each project hospital and 37 other hospitals based on the principle of voluntary participation. A total of 328 hospitals completed information collection.

This project will establish standards for nutrition risk assessment, diagnosis, and treatment of inpatients in China, promote the construction of clinical nutrition departments, and improve the nutritional status of inpatients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Admitted to hospital within 24-48 hours (not emergency) due to tumor or digestive system, respiratory system, cardiovascular system, endocrine system, nervous system, and urinary system disease.

Exclusion Criteria:

* With mental illness or memory disorder who were unable to answer questions correctly
* Critically ill patients
* Lack behavioral ability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A large, nationally representative sample of Chinese adult inpatients
Sampling Method: Probability Sample
Enrollment: 54677 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Number of participants diagnosed with malnutrition | The 1 day of the survey
  For the diagnosis of malnutrition, we adopted the Global Leadership Initiative on Malnutrition (GLIM) scheme based on three phenotypic criteria (non-volitional weight loss, low body mass index, and reduced muscle mass) and two etiologic criteria (reduced food intake or assimilation, and inflammation or disease burden). To diagnose malnutrition at least one phenotypic criterion and one etiologic criterion should be present in patients with nutritional risk.
Prevalence of nutritional risk | The 1 day of the survey
  Nutritional risk was defined as Nutritional Risk Screening 2002 (NRS2002) score≥3.

CONTACTS AND LOCATIONS:
Locations (1):
- Dongcheng district，Peking union medical college hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Deng LM, Liu SP, Long JF, Mo H, Liu M, Liu JY, Zhang YL, Xu DF, Yu HZ, Chen L, Cai H, Yang SB, Xiang M, Liu M, Sun Y, Xie ZJ, Zeng MM, Xie GX. Prevalence of malnutrition and appropriateness of nutritional support in hospitalized patients: a GLIM-based study. Front Nutr. 2025 Oct 10;12:1667821. doi: 10.3389/fnut.2025.1667821. eCollection 2025. PMID 41141257